CLINICAL TRIAL: NCT06429683
Title: Effectıveness of The Sexually Transmıtted Dıseases Educatıon Program for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahar Nur Kanbur (Other)
Responsible Party: Sponsor-Investigator, Bahar Nur Kanbur, Assistant Professor, Istanbul Gelisim University
Organization: Istanbul Gelisim University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IstanbulGelisimuniversity
Record Dates: First submitted 2024-05-17; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Sexually Transmitted Diseases
Keywords: adolescent; sexually transmitted diseases; education
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sexually transmitted diseases training for young adolescents aged 17-21 (Experimental): To evaluate the effectiveness of sexually transmitted diseases education given to young adolescents aged 17-21 years
  Interventions: Other: Sexually transmitted diseases training for young adolescents aged 17-21

INTERVENTIONS:
Other: Sexually transmitted diseases training for young adolescents aged 17-21 — Education

SUMMARY:
The World Health Organization has defined the period between the ages of 10-19 as adolescence, 15-24 years as youth and 10-24 years as youth period. Adolescence is divided into 3 periods: early adolescence (10-13 years), middle adolescence (14-16 years) and late adolescence (17-21 years). HIV virus and AIDS, which have become a problem among sexually transmitted diseases all over the world, have increased the importance of controlling sexually transmitted diseases. There is a strong correlation between the spread of STDs through traditional means and the transmission of HIV; and sexually transmitted diseases have been found to increase the risk of sexual transmission of HIV. According to WHO data, 340 million treatable STDs, millions of incurable STDs and 5 million HIV cases occur worldwide each year.

DETAILED DESCRIPTION:
People in the 15-49 age group who are sexually active are the most likely to contract sexually transmitted diseases. The prevalence of STDs is higher in developing countries than in developed countries. These diseases are among the top 5 etiologic factors that cause loss of years of "healthy productive life" in developing countries. As in other countries, sexually transmitted diseases are of great importance in terms of complications and sequelae in Turkey

One out of 20 young people is infected with STDs every year. In our country, the age of sexual maturation has shifted earlier. In addition, the age of sexual experience of young people has also shifted earlier. Young people's understanding of freedom and their inability to access FP methods whenever they want negatively affect their sexual health behaviors. Impact on Society STDs cause a lot of economic and social damage to society. STDs may disrupt the normal functioning of family, community and health institutions and leave these institutions under a heavy economic burden. STDs reduce the productivity of men and women at the most productive ages of their lives. In addition, when outbreaks of these infections are not controlled, the costs to society will increase.

Translated with DeepL.com (free version)

ELIGIBILITY:
Inclusion Criteria:

* At a Foundation University located within the borders of Istanbul Province 1.2.3. and 4th grade students

Exclusion Criteria:

-

Ages: 17 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 250 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Students' Knowledge Test on Sexually Transmitted Diseases | 2 months
  The Sexually Transmitted Diseases Knowledge Test includes 36 questions that assess students' level of knowledge about sexually transmitted diseases. The questions are answered as "True", "False", and "I don't know". Students will be administered the STD knowledge test before the training. The test will be administered again after the training. In the post-training test, the student is expected to give more correct answers to the questions compared to the previous test.

CONTACTS AND LOCATIONS:
Overall Officials: Canan Örüklü, Principal Investigator — Trakya University
Locations (1):
- Istanbul Gelisim University, Istanbul, Avcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No